CLINICAL TRIAL: NCT06459622
Title: Predictive Factors in Chronic Rhinosinusitis With Nasal Polyps
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Katrina Atef Habashy (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Katrina Atef Habashy, Predictive factors in response of chronic rhinosinusitis with nasal polyps to corticosteroids, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: Chronic rhinosinusitis
Record Dates: First submitted 2024-03-31; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-03

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensitive to corticosteroids (Experimental): Patients who are sensitive to corticosteroids have high serum IL-25
  Interventions: Diagnostic Test: Serum IL_25 and eosinophils in nasal polyp tisuee
- Non sensitive to corticosteroids (Experimental): Patients who aren't sensitive to corticosteroids have low serum IL-25
  Interventions: Diagnostic Test: Serum IL_25 and eosinophils in nasal polyp tisuee

INTERVENTIONS:
Diagnostic Test: Serum IL_25 and eosinophils in nasal polyp tisuee — Serum IL-25 and eosinophils in nasal polyps tisuer obtained and measured to identify the sensitivity of nasal polyps to corticosteroids

SUMMARY:
The study will be conducted to identify factors predicting the response of chronic rhinosinusitis with nasal polyps ( CRSwNP) to oral corticosteroids.

DETAILED DESCRIPTION:
Treatment of nasal polyposis is divided into medical or surgical treatment .

Steroids are widely used as the most effective medicine in nasal polyposis. Although oral corticosteroids are one of the frequently used treatments in the management of chronic rhinosinusitis with nasal polyps (CRSwNP), there is lack of effective means of predicting corticosteroid sensitivity in those patients. It was reported that the overall sensitivity rates of corticosteroid therapy to nasal polyps( NP) were only between 53.8% and 80%.. Many reports stated that serum and tissue interleukeine 25 (IL 25) and serum and tissue eosinophalia are good predictors to the response of CRSwNP to oral corticosteroids.

Interleukeine 25(IL-25), an important epithelial-derived proinflammatory cytokine, plays various roles in different inflammatory and allergic diseases, such as asthma and atopic dermatitis .

Hong et al demonstrated that the levels of IL-25 in NP tissues and in serum, as well as the NP endoscopic scores, were significantly elevated in the corticosteroid-sensitive patients compared with the non-sensitive ones. In general, eosinophilic NPs are pharmacologically glucocorticoid responsive, but non-eosinophilic or neutrophilic CRSwNP is frequently resistant to steroid treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of chronic rhinosinusitis with nasal polyps

Exclusion Criteria:

* 1-Patients who had taken any steroid , antihistamine or other immune-modulating medications within the past 4 weeks

  2- previous nasal and sinus surgery.

  3-Allergic Fungal rhinosinusitis.

  4-Unilateral rhinosinusitis.

  5- Antrochoanal polyps or cystic fibrosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Serum IL-25 is measured to releave the relation between them and the response of CRSwNP to oral corticosteroids | Baseline
  Serum IL-25 is related to the effect of corticosteroids on CRSwNP

OTHER OUTCOMES:
Eosinophils in nasal polyp tissue | Baseline
  Eosinophils is related to the inflammatory process of CRSwNP

REFERENCES:
- [Background] Shin HW, Kim DK, Park MH, Eun KM, Lee M, So D, Kong IG, Mo JH, Yang MS, Jin HR, Park JW, Kim DW. IL-25 as a novel therapeutic target in nasal polyps of patients with chronic rhinosinusitis. J Allergy Clin Immunol. 2015 Jun;135(6):1476-85.e7. doi: 10.1016/j.jaci.2015.01.003. Epub 2015 Feb 25. PMID 25725991
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/29337030/